CLINICAL TRIAL: NCT02970734
Title: Evaluating an Internet-based Program for Anxious Adolescents: A Randomized Controlled Trial
Brief Title: Evaluating an Internet-based Program for Anxious Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00066393
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2018-09

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breathe (Experimental): 6 sessions of Internet-based cognitive behavioural therapy (CBT) with limited telephone and e-mail support
  Interventions: Behavioral: Breathe
- Resource webpage (Active Comparator): Webpage that provides general resources on anxiety
  Interventions: Behavioral: Resource Webpage

INTERVENTIONS:
Behavioral: Breathe — Six web-based cognitive behavioural therapy sessions. Telephone and email support are also provided during the program.
  Arms: Breathe
Behavioral: Resource Webpage — Static webpage listing anxiety resources.
  Arms: Resource webpage

SUMMARY:
Anxiety is a common mental health problem for Canadian adolescents. Anxiety that is diagnosed as a disorder and serious enough to require treatment affects up to 10% of all adolescents by the age of 16. The median age of onset is 11 years, making these disorders some of the earliest to develop. Anxiety disorders can have serious negative effects on a young person's personal relationships, school performance, and family life. These disorders may not be discovered by adolescents, parents and health care providers. Even if anxiety disorders are discovered, adolescents may not get the right therapy. Anxious adolescents can become sick if their anxiety is not treated properly. The investigators will carry out research to test Breathe, an Internet-based treatment for adolescents with anxiety problems. Adolescents can use this treatment from home via the computer. Breathe will include information materials and personalized homework assignments to help anxious adolescents learn ways to manage anxiety. More information can be found and www.TheBreatheStudy.com

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) with two groups, an Internet-delivered cognitive behavioural therapy (CBT) experimental group (Breathe) and a resource webpage (control group; considered treatment as usual for youth waiting for services). The investigators will evaluate several methodological processes and outcomes through the following objectives:

1. To determine the effectiveness of a self-guided Internet-based CBT program with limited telephone and email support in reducing anxiety symptoms among adolescents with mild-to-moderate anxiety as compared to a usual self-help intervention, a resource-based webpage.
2. To explore mediators and moderators of the Internet-based CBT program.
3. To determine the effectiveness of a self-guided Internet-based CBT program in improving quality of life as compared to a usual self-help intervention.
4. To determine adherence to a self-guided Internet-based CBT program.
5. To determine the cost-effectiveness of the Internet-based CBT program.

ELIGIBILITY:
Inclusion Criteria:

* Score of ≥25 on the Screen for Child Anxiety Related Disorders (SCARED)
* Ability to read and write English
* Regular access to a telephone and a computer system with high speed Internet service
* Ability to use the computer to interact with web material

Exclusion Criteria:

* Positive screen on the Ask Suicide-Screening Questionnaire (ASQ)
* Positive screen on the Schizophrenia Test and Early Psychosis Indicator (STEPI; modified version)
* Score of ≥3 on the Alcohol Use Disorders Identification Test Consumption subscale (AUDIT-C)
* Residence outside of Canada

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 563 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Change in adolescent anxiety using the total Multidimensional Anxiety Scale for Children (MASC 2) score | baseline to 6 weeks post-baseline (post-intervention)

SECONDARY OUTCOMES:
Change in adolescent anxiety using the total MASC 2 score | 6 weeks post-baseline (post-intervention) to 18 weeks post-baseline (3-month follow-up)
Change in quality of life using the Youth Quality of Life Instrument - Short Form (YQOL-SF) | baseline to 6 weeks post-baseline (post-intervention), 6 weeks post-baseline (post-intervention) to 18 weeks post-baseline (3-month follow-up)
User experience | 6 weeks post-baseline (post-intervention)
  Developed by the investigators, this electronically administered, self-report instrument will assess participant satisfaction (e.g., ease of use, layout, convenience) perceived credibility and impact (e.g., helpfulness, knowledge gains, confidence in the program/website), and adherence and usage (e.g., barriers and facilitators to treatment) with an Internet-based program/webpage.
Intervention adherence | 6 weeks post-baseline (post-intervention)
  Intervention adherence will be measured by documenting the number of sessions and homework tasks completed. The investigators will also record the number of tailored sessions completed by each participant (intervention condition) and site visits (control condition). These data will be collected through the intervention's software system.
health care utilization | baseline, 18 weeks post-baseline
  Developed by the investigators, this self-report instrument will assess whether participants have accessed health care resources (i.e., met with a psychologist/psychiatrist/family doctor/hospital etc.) and if so, how many times.

OTHER OUTCOMES:
Recruitment rate | Through study conduct, an average of 1 year.
Retention rate | Through study conduct, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Newton, Principal Investigator — University of Alberta
Locations (1):
- The Breathe Team, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connor KA, Bagnell A, Rosychuk RJ, Chen AA, Lingley-Pottie P, Radomski AD, Ohinmaa A, Joyce A, McGrath PJ, Newton AS. A randomized controlled trial evaluating the effect of an internet-based cognitive-behavioral program on anxiety symptoms in a community-based sample of adolescents. J Anxiety Disord. 2022 Dec;92:102637. doi: 10.1016/j.janxdis.2022.102637. Epub 2022 Sep 24. PMID 36179438
- [Derived] Radomski AD, Bagnell A, Curtis S, Hartling L, Newton AS. Examining the Usage, User Experience, and Perceived Impact of an Internet-Based Cognitive Behavioral Therapy Program for Adolescents With Anxiety: Randomized Controlled Trial. JMIR Ment Health. 2020 Feb 7;7(2):e15795. doi: 10.2196/15795. PMID 32022692